CLINICAL TRIAL: NCT06547216
Title: A Phase 2 Open-label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of AOC 1020 Administered Intravenously to Participants with Facioscapulohumeral Muscular Dystrophy (FSHD)
Brief Title: Phase 2 Open-label Extension Study of AOC 1020 in Participants with Facioscapulohumeral Muscular Dystrophy (FSHD)
Acronym: FORTITUDE-OLE
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Avidity Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOC 1020-CS2
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: FSHD; FSHD1; FSHD2; FMD; FMD2; Fascioscapulohumeral Muscular Dystrophy; Fascioscapulohumeral Muscular Dystrophy Type 1; Fascioscapulohumeral Muscular Dystrophy Type 2; Dystrophies, Facioscapulohumeral Muscular; Dystrophy, Facioscapulohumeral Muscular; Facioscapulohumeral Muscular Dystrophy 1; Facioscapulohumeral Muscular Dystrophy 2; Facio-Scapulo-Humeral Dystrophy; Atrophy, Facioscapulohumeral; Atrophies, Facioscapulohumeral; Facioscapulohumeral Atrophy; Muscular Dystrophies; Muscular Dystrophy, Facioscapulohumeral; FSH Muscular Dystrophy; Landouzy Dejerine Dystrophy; Landouzy-Dejerine Muscular Dystrophy; Dystrophies, Landouzy-Dejerine; Dystrophy, Landouzy-Dejerine; Landouzy-Dejerine Syndrome; Muscular Dystrophy, Landouzy Dejerine; Progressive Muscular Dystrophy; FSH
Keywords: FORTITUDE; Avidity; Avidity Biosciences; AOC 1020; FORTITUDE-OLE; FORTITUDE OLE
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Facioscapulohumeral Muscular Dystrophy 1B; Muscular Dystrophies; Facioscapulohumeral muscular dystrophy 1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AOC 1020 Regimen (Experimental): AOC 1020 Dose Regimen; Sixteen doses administered intravenously over 22 months. All participants will receive AOC 1020 at a dose level of 2mg/kg.
  Interventions: Drug: AOC 1020

INTERVENTIONS:
Drug: AOC 1020 — AOC 1020 will be administered via intravenous (IV) infusion
  Other Names: delpacibart braxlosiran; del-brax

SUMMARY:
A Phase 2 Open-label Extension Study to Evaluate the Long-Term Safety, Tolerability, and Efficacy of AOC 1020 Administered Intravenously to Participants with Facioscapulohumeral Muscular Dystrophy (FSHD)

DETAILED DESCRIPTION:
This study will continue to evaluate the safety, tolerability, and efficacy of AOC 1020 in participants who were treated in the randomized, placebo-controlled, Phase 1/2 AOC 1020-CS1 clinical study.

Participants from AOC 1020-CS1 are eligible to enroll in AOC 1020-CS2 if they have satisfactorily completed AOC 1020-CS1. All participants who enroll in AOC 1020-CS2 will receive AOC 1020 regardless of whether they received AOC 1020 or placebo in AOC 1020-CS1. Dosing will occur every 6 to 7 weeks (twice quarterly).

The total duration of active treatment in AOC 1020-CS2 is approximately 22 months. Once participants have completed active treatment, they will be followed through a 12-week safety follow-up period to monitor for adverse events (AEs), concomitant medications, and pregnancy status (as applicable). Total duration on study is up to approximately 25 months (2 years 1 month), excluding the potential 8-week screening period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent (signed and dated) and any authorizations required by local law and be willing and able to comply with all study requirements. When enrolling participants who are minors, it is necessary to also obtain consent from a legally designated representative and the participant will receive information in a way adapted to their age and mental maturity.
2. Completion of AOC 1020-CS1 with the following as judged by the Investigator and Sponsor:

   1. No significant tolerability issues
   2. Satisfactory compliance with the AOC 1020-CS1 protocol requirements

Exclusion Criteria:

1. Pregnancy, intent to become pregnant during the clinical study, or active breastfeeding.
2. Unwilling or unable to continue to comply with contraceptive requirements for the length of AOC 1020-CS2.
3. Any new conditions or worsening of existing condition(s) that in the opinion of the Investigator or Sponsor would make the participant unsuitable for the study or could interfere with participation or completion of the study. (Note: FSHD progression is not exclusionary, even if the participant no longer has the ability to walk 10 meters without a walker or two canes.)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Through study completion, up to Day 729

CONTACTS AND LOCATIONS:
Overall Officials: Amy Halseth, Ph.D., Study Director — Avidity Biosciences, Inc.
Locations (17):
- United States (14):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California San Diego, San Diego, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Rare Disease Research, Atlanta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Rochester Medical Center, Rochester, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- University of Ottawa, Ottawa, Ontario, Canada
- United Kingdom (2):
  - University College London, London
  - University of Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Avidity Biosciences Website — https://www.aviditybiosciences.com/